CLINICAL TRIAL: NCT02012881
Title: LCoMotion. Learning, Cognition and Motion. Effect of a Four Month School-based Cluster-randomized Intervention
Acronym: LCoMotion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Ministry of Education, Denmark (Other Government)
Responsible Party: Principal Investigator, Anna Bugge, Post Doc, Post Doc, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S-20130104
Record Dates: First submitted 2013-10-11; First posted 2013-12-16 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Cognitive Function

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical activity intervention (Experimental): 60 minutes of physical activity on every school day
  Interventions: Behavioral: Physical activity intervention
- Control (Active Comparator): Usual practice
  Interventions: Behavioral: Usual practice

INTERVENTIONS:
Behavioral: Physical activity intervention — Physical activity during recess, in academic subjects, active transportation and PA home work
  Arms: Physical activity intervention
Behavioral: Usual practice — Normal curriculum
  Arms: Control

SUMMARY:
The purpose of this study is to determine the effect of a four months school-based physical activity intervention on cognition, academic achievement, physical activity and aerobic fitness in 12-15 year old adolescents.

ELIGIBILITY:
Inclusion Criteria:

* six or seventh grader in a Danish public school
* participating in normal math lessons

Exclusion Criteria:

* private school
* receiving extra math lessons because of special needs

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 870 (Actual)
Dates: Start 2013-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Executive function accuracy | Up to 8 months
  Executive function (part of cognitive function) measured by a modified computer-based flanker-test

SECONDARY OUTCOMES:
Academic achievement | November 2013 -June 2014
  A standardized math test
Physical activity | November 2013-June 2014
  Measured with accelerometers for one week both pre- and post-intervention and supplemented with a questionnaire
Aerobic fitness | November 2013 - June 2014
  Measured with an intermittent running test (Andersen test)
Anthropometric measures | November 2013 - June 2014
  Body height, body weight, waist circumference and puberty status (self-assessed)
Questionnaire | November 2013 - June 2014
  To students and parents. SES, family diseases, physical activity, sport participation

OTHER OUTCOMES:
SMS tracking | November 2013- June 2014
  Asking questions on compliance with the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Sports Science and Clinical Biomechanics, Odense, Denmark

REFERENCES:
- [Derived] Tarp J, Domazet SL, Froberg K, Hillman CH, Andersen LB, Bugge A. Effectiveness of a School-Based Physical Activity Intervention on Cognitive Performance in Danish Adolescents: LCoMotion-Learning, Cognition and Motion - A Cluster Randomized Controlled Trial. PLoS One. 2016 Jun 24;11(6):e0158087. doi: 10.1371/journal.pone.0158087. eCollection 2016. PMID 27341346
- [Derived] Bugge A, Tarp J, Ostergaard L, Domazet SL, Andersen LB, Froberg K. LCoMotion - Learning, Cognition and Motion; a multicomponent cluster randomized school-based intervention aimed at increasing learning and cognition - rationale, design and methods. BMC Public Health. 2014 Sep 18;14:967. doi: 10.1186/1471-2458-14-967. PMID 25236478